CLINICAL TRIAL: NCT04520893
Title: Modification of Ventilation Strategy for the Elderly Patients During Spine Surgery in Prone Position
Brief Title: Ventilation Strategy for the Elderly Patients in Prone Position
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Eunhee Chun (Other)
Responsible Party: Sponsor-Investigator, Eunhee Chun, Assistant professor, Hallym University Kangnam Sacred Heart Hospital
Organization: Hallym University Kangnam Sacred Heart Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-03-010
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Ventilators, Mechanical
Keywords: geriatric medicine, protective ventilation, prone position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VCV pause (Experimental): volume controlled ventilation with pause time 30%
  Interventions: Procedure: ventilator setting vcv with pause
- VCV (Active Comparator): volume controlled ventilation (without pause)
  Interventions: Procedure: ventilator setting vcv
- PCV-VG (Active Comparator): pressure controlled ventilation - volume guaranteed
  Interventions: Procedure: ventilator setting pcv-vg

INTERVENTIONS:
Procedure: ventilator setting vcv with pause — ventilator setting vcv with pause
  Arms: VCV pause
Procedure: ventilator setting vcv — ventilator setting vcv without pause
  Arms: VCV
Procedure: ventilator setting pcv-vg — ventilator setting with pcv-vg
  Arms: PCV-VG

SUMMARY:
The investigators compare three ventilation modes; volume controlled ventilation, volume guaranteed pressure controlled ventilation and volume controlled ventilation with pause during spine surgery for the elderly patients. The investigators can reveal that how lung collapse can be reduced by optimizing the inspiratory flow pattern under general anesthesia.

DETAILED DESCRIPTION:
<Protocol>

1. All patients were ventilated by an anaesthesia ventilator (Zeus, Dräger, Lübeck, Germany) under general anesthesia.
2. Ventilation strategy:

   * Pressure controlled ventilation volume guaranteed (PCV-VG) mode or volume control ventilation (VCV) mode
   * tidal volume 6-8 mL/kg (predicted body weight)
   * Inspiratory/expiratory (I/E) ratio 1:1.5
   * Inspired oxygen concentration (FIO2) 0.5 with air
   * 3.0 L/min of inspiratory fresh gas flow
   * Positive end-expiratory pressure (PEEP) of 5 cm H2O
   * Respiratory rate (RR) of 10 to 14 min-1
3. After prone positioning and hemodynamic condition was stabilized, patients were ventilated with VCV, PCV-VG mode, VCV with pause following a randomized order, previously determined for each patient. Before each ventilator setting was started, lung recruitment maneuvers were performed to set the lungs to a defined baseline status.

   * ventilation order : one of the following examples is taken by randomization.

VCV 15 min -- VCV pause 15min -- PCV-VG 15min

VCV 15 min -- PCV-VG 15min -- VCV pause 15min

VCV pause 15min -- VCV 15 min -- PCV-VG 15min

VCV pause 15min -- PCV-VG 15min -- VCV 15 min

PCV-VG 15min -- VCV 15 min -- VCV pause 15min

PCV-VG 15min -- VCV pause 15min -- VCV 15 min

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective spine surgery under general anesthesia

Exclusion Criteria:

* obesity (body mass index >35 kg/m2)
* chronic obstructive pulmonary disease
* respiratory infection

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
MVCO2 | ventilation 15 min later
  minute CO2 production (ml/min), a parameter of Drager ventilator, displayed in the Primus model and software

SECONDARY OUTCOMES:
airway pressure | ventilation 15 min later
  peak airway pressure (cmH2O; displayed in the ventilator), plateau pressure (cmH2O; diaplayed in the ventilator), driving pressure(cmH2O, plateau pressure minus peak airway pressure)
airway compliance | ventilation 15 min later
  Respiratory dynamic compliance (ml/cmH2O; displayed in the ventilator)

CONTACTS AND LOCATIONS:
Overall Officials: Eunhee Chun, MD.,PhD., Principal Investigator — Hallym University Kangnam Sacred Heart Hospital
Locations (1):
- Hallym University Kangnam Sacred Hospital, Seoul, South Korea